CLINICAL TRIAL: NCT06918405
Title: Efficacy and Safety of Tirzepatide for Weight Management in Overweight or Obese Adult Individuals With or Without Type 2 Diabetes Mellitus: A Real-World Study in Bangladesh
Brief Title: Efficacy and Safety of Tirzepatide for Weight Management
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Dr. Fahmida Islam Chowdhury, Associate Professor, Chittagong Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59.127.1557.013.19.PG.2025/337
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Obesity; Tirzepatide; Type 2 diabetes mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide arm (Experimental): All the included patients in both the diabetic and nondiabetic groups will receive the same intervention of tirzepatide at a dose of 15 mg administered subcutaneously once a week in addition to lifestyle modification.
  Initially, tirzepatide will be started with a dose of 2.5 mg once weekly subcutaneous injection for the first 4 weeks. After the stabilization period of the drug, the dose will be increased to 5 mg after 4 weeks, 7.5 mg after 8 weeks, 10 mg after 12 weeks, 12.5 mg after 16 weeks and finally 15 mg after 20 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — All the included patients in both the diabetic and nondiabetic groups will receive the same intervention of tirzepatide at a dose of 15 mg administered subcutaneously once a week in addition to lifestyle modification.
  Initially, tirzepatide will be started with a dose of 2.5 mg once weekly subcutaneous injection for the first 4 weeks. After the stabilization period of the drug, the dose will be increased to 5 mg after 4 weeks, 7.5 mg after 8 weeks, 10 mg after 12 weeks, 12.5 mg after 16 weeks and finally 15 mg after 20 weeks.

SUMMARY:
The goal of this study is to learn if tirzepatide helps people manage their weight safely. It will include adults in Bangladesh who are overweight or obese, with or without type 2 diabetes. The main questions it aims to answer are:

Does tirzepatide help people lose weight?

What side effects do people experience while taking tirzepatide?

All participants will:

Receive tirzepatide as a weekly injection, starting at 2.5 mg and gradually increasing to 15 mg.

Continue the treatment for 52 weeks (12 months).

Visit the clinic for regular checkups and tests.

Researchers will measure changes in body weight, BMI, waist size, blood sugar, blood pressure, and cholesterol levels. They will also track any side effects and assess the participants' overall health and quality of life during the study.

DETAILED DESCRIPTION:
Obesity has emerged as a critical global public health issue, significantly linked to an increased risk of various comorbidities, including type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, and cardiovascular diseases. While lifestyle modifications, such as adhering to a low-calorie diet and enhancing physical activity, remain the cornerstone of obesity management, the recent development of anti-obesity medications such as GLP-1 agonists has transformed treatment options. This study aims to evaluate the efficacy and safety of tirzepatide, GLP-1 agonist, in weight management among overweight or obese adult individuals, both with and without T2DM in Bangladesh.

This single treatment arm clinical trial will be conducted in a real-world setting, enrolling male and female adults aged 18 years or older, with a body mass index (BMI) of ≥30 kg/m² or ≥25-29.9 kg/m² if they have at least one weight-related comorbidity, such as, hypertension, or dyslipidemia. All the individuals recruited in the present study will receive subcutaneous injections of tirzepatide, initiated at a dose of 2.5 mg once weekly for the first four weeks, with incremental increases of 2.5 mg every four weeks, reaching the maintenance dose of 15 mg once weekly. The follow-up period will be 52 weeks (12 months) from the start of treatment.

The primary efficacy endpoint will be the percentage change in body weight from baseline at week 52. Secondary endpoints will include the proportion of participants achieving weight reductions of ≥5%, ≥10%, ≥15%, and ≥20% after 52 weeks, as well as changes in body weight (kg), BMI (kg/m²), waist circumference (cm), HbA1c (%), fasting plasma glucose (FPG) (mg/dL), blood pressure (both systolic and diastolic), serum lipid levels (mg/dL), modifications in hypoglycemic and antihypertensive medications, and overall quality of life assessed through an obesity-specific QoL instrument. The study will also evaluate the incidence and severity of adverse events, alongside physical examination results, blood pressure measurements, and laboratory parameter changes from baseline.

Adhering to Good Clinical Practice Guidelines, this study will follow ethical principles outlined in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria

Common inclusion criteria for both diabetic and non-diabetic individuals:

* Informed consent will be obtained before any trial-related activities.
* Male or female, aged ≥18 years at the time of signing the informed consent form.
* Have a history of at least one self-reported unsuccessful dietary effort to lose body weight.
* Body mass index (BMI):
* ≥30 kg/m² with or without any weight-related comorbidities or
* ≥25-29.9 kg/m² with the presence of at least one of the following weight-related comorbidities (treated or untreated):
* Hypertension (systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg or currently taking antihypertensive medication).
* Dyslipidemia (treated or with low-density lipoprotein (LDL) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein (HDL) <40 mg/dL (1.0 mmol/L) for men or HDL <50 mg/dL (1.3 mmol/L) for women).
* Obstructive sleep apnea.
* Cardiovascular disease (more than three months).
* In the investigator's opinion, are well-motivated, capable, and willing to:
* Learn how to self-inject study drug, as required for this protocol (visually impaired persons who are not able to perform the injections must have the assistance of a sighted individual trained to inject study drug; persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject study drug).
* Inject study drug (or receive an injection from a trained individual if visually impaired or with physical limitations).
* Follow study procedures for the duration of the study, including, but not limited to, following lifestyle advice (for example, dietary restrictions and exercise plan) and maintaining a study diary.
* Male participants:
* Male participants with partners of childbearing potential should be willing to use reliable contraceptive methods throughout the study and for 5 half-lives of the study drug plus 90 days, corresponding to 4 months after the last injection.
* Female participants:
* Female participants not of childbearing potential may participate and include those who are:
* Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenesis.
* Postmenopausal, defined as either:
* A woman at least 40 years of age with an intact uterus, not on hormone therapy, who has cessation of menses for at least 1 year without an alternative medical cause, AND a follicle-stimulating hormone ≥40 mIU/mL; women in this category must test negative in pregnancy test prior to study entry.
* A woman 55 or older not on hormone therapy, who has had at least 12 months of spontaneous amenorrhea.
* A woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy.
* Female participants of childbearing potential (not surgically sterilized and between menarche and 1-year postmenopausal) must:
* Test negative for pregnancy at Visit 1 based on a serum pregnancy test.
* If sexually active, agree to use 2 forms of effective contraception, where at least 1 form is highly effective, for the duration of the trial and for 30 days thereafter.
* Not be breastfeeding.

For subjects with T2DM:

* Patients diagnosed with T2DM more than or equal to 180 days prior to the day of screening.
* HbA1c up to 10.0%.

Exclusion Criteria

Common exclusion criteria for both diabetic and non-diabetic individuals:

* Medical criteria:
* Have obesity induced by other endocrinologic disorders (for example, Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome).
* A self-reported reduction in body weight of more than 5 kg within 30 days before screening, irrespective of medical records.
* Treatment with any medication for the indication of obesity within the past 90 days before screening (e.g., Orlistat, liraglutide, naltrexone/bupropion, diethylpropion, phendimetrazine, semaglutide, and setmelanotide).
* Any previous obesity treatment with surgery or a weight loss device during a lifetime.
* Continued treatment with other GLP-1 agonists, SGLT-2 inhibitors, and/or metformin. However, if these drugs can be stopped based on the best clinical judgment of the investigator, the patient can be recruited after stopping the drug and a washout period of two weeks. In the case of tirzepatide, the washout period will be 8 weeks.
* Are receiving or have received within 3 months prior to screening chronic (>2 weeks or 14 days) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, intra-articular, or inhaled preparations) or have evidence of a significant, active autoimmune abnormality (for example, lupus or rheumatoid arthritis).
* Have current or history of (within 3 months prior to enrollment) treatment with medications that may cause significant weight gain, including but not limited to tricyclic antidepressants, atypical antipsychotics, and mood stabilizers.
* Have started implantable or injectable contraceptives (such as Depo-Provera®) within 18 months prior to screening.
* Past history of pancreatitis.
* Diagnosed case of eating disorders (e.g., Bulimia nervosa).
* Patients with a previous history of suicide attempts and major depressive disorder (MDD) according to DSM-V criteria, schizophrenia, or antipsychotic drug-induced obesity.
* Patients with a personal or family history of medullary thyroid carcinoma (MTC) and/or multiple endocrine neoplasia syndrome type 2 (MEN 2).
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years.
* Have uncontrolled hypertension (SBP ≥160 mmHg and/or DBP ≥100 mmHg).
* Have NYHA Functional Classification IV CHF.
* Have had a transplanted organ (corneal transplants [keratoplasty] allowed) or awaiting an organ transplant.
* Laboratory criteria:
* Incidental diagnosis or uncontrolled thyroid disease, defined as a thyroid-stimulating hormone (TSH) level >6.0 mIU/L or <0.4 mIU/L as measured by the central laboratory at screening. However, well-controlled thyroid disorder can be included if TSH <6.0 or >0.4 mIU/L.
* Renal impairment, measured as the estimated glomerular filtration rate (eGFR) <15 ml/min/1.73 m².

For subjects without T2DM:

- HbA1c more than or equal to 48 mmol/mol (6.5%).

For subjects with T2DM:

* Renal impairment, defined as an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73 m² (less than 60 mL/min/1.73 m² in subjects treated with a sodium-glucose cotransporter 2 inhibitor (SGLT2i)).
* Uncontrolled T2DM (HbA1c >10.0%) as these patients may require insulin or other anti-diabetic drugs which might potentially interfere with the efficacy of tirzepatide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight (kg) | 52 weeks
  Change in body weight (kg) [5%, 10%, 15% and 20%] from baseline at week 0 to week 52

SECONDARY OUTCOMES:
Change in BMI | 52 weeks
  Change in BMI (kg/m2) from baseline at week 0 to week 52
Change in Waist circumference | 52 weeks
  Change in Waist circumference (cm) from baseline at week 0 to week 52
Change in HbA1c | 52 weeks
  Change in HbA1c (%) from baseline at week 0 to week 52
Change in fasting plasma glucose | 52 weeks
  Change in fasting plasma glucose (FPG) (mg/dl) from baseline at week 0 to week 52
Change in blood pressure | 52 weeks
  Change in systolic and diastolic blood pressure (mmHg) from baseline at week 0 to week 52
Change in lipid profile | 52 weeks
  Change in lipid profile (mg/dl) from baseline at week 0 to week 52 i. Total cholesterol ii. High-density lipoprotein (HDL) cholesterol iii. Low-density lipoprotein (LDL) cholesterol iv. Triglycerides
Change in serum creatinine | 52 weeks
  Change in serum creatinine (mg/dl) from baseline at week 0 to week 52
Dose alteration in antidiabetic drugs | 52 weeks
  Dose alteration (reduction or increment) or change/addition of hypoglycemic agents in patients with T2DM from baseline at week 0 to week 52
Dose alteration of antihypertensive drugs | 52 weeks
  Dose alteration (reduction or increment) or change/addition of antihypertensive agents in patients with hypertension from baseline at week 0 to week 52
Change in quality of life | 52 weeks
  Patients' overall quality of life, measured by the Obesity-specific QoL instrument (OSQOL). The instrument includes four domains: physical state, vitality, social interactions, and psychological state
Adverse events | 52 weeks
  Number of treatment-related adverse events and serious adverse events (SAEs) from baseline at week 0 to week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided